CLINICAL TRIAL: NCT03437902
Title: Evaluation of the Impact of Rutin and Vitamin C Combination on Oxidative Stress, Insulin Sensitivity and Lipid Profile in Type 2 Diabetic Patients
Brief Title: Impact of Rutin and Vitamin C Combination on Oxidative Stress, Insulin Sensitivity and Lipid Profile in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, sara ramzy ragheb, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL39
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; Rutin; Vitamin C; oxidative stress; Insulin resistance; lipid profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Rutin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rutin C group (Experimental): patients will receive Rutin 60 mg in combination with vitamin C 160 mg three times daily in addition to usual antidiabetic treatment for 8 weeks..
  Interventions: Dietary Supplement: Rutin in combination with Vitamin C
- Vitamin C group (Experimental): patients will receive vitamin C 500 mg once daily in addition to usual antidiabetic treatment for 8 weeks.
  Interventions: Dietary Supplement: Vitamin C
- Control group (No Intervention): patients will receive their usual antidiabetic treatment only for 8 weeks.

INTERVENTIONS:
Dietary Supplement: Rutin in combination with Vitamin C — Rutin and Vitamin C will be supplied as tablets containing 60 mg Rutin and 160 mg Vitamin C. The use of Rutin and Vitamin C will be under the trade name of RUTA C 60 ® manufactured by KAHIRA PHARM.& CHEM. IND. Company
  Arms: Rutin C group
Dietary Supplement: Vitamin C — Vitamin C will be supplied as capsules containing500 mg of Vitamin C. The use of Vitamin C will be under the trade name of C-Retard ® manufactured by HIKMA Quality Company.
  Other Names: Ascorbic acid
  Arms: Vitamin C group

SUMMARY:
The objective of this study is to investigate the effect ofRutin and Vitamin C combination in comparison with vitamin C alone on the oxidative and antioxidative status , insulin resistance and lipid profile in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* • Patients' age 35 years or older having type 2 diabetes mellitus.

  * Patients taking oral diabetic medications (Sulfonylurea) not taking Insulin.
  * Able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* • Pregnant and breast feeding females

  • use of vitamin supplements containing vitamin C or other antioxidants.
* patients with renal or hepatic failure.
* patients taking insulin as antidiabetic treatment

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Oxidative stress marker (MDA) and antioxidant capacity (SOD) in diabetic patients | Two months
  Effect of Rutin and vitamin C combination or vitamin C alone on oxidative stress marker (MDA) and on antioxidant capacity (SOD) in diabetic patients after 8 weeks of treatment.
Insulin resistance in diabetic patients . | Two months
  Effect of Rutin and vitamin C combination or vitamin C alone on insulin resistance in diabetic patients before i and after treatment for 8 weeks .
Lipid profile in diabetic patients (TC,TG,HDL-c,LDL-c). | Two months
  Impact of Rutin and vitamin C combination or vitamin C alone on lipid profile in diabetic patients (TC,TG,HDL-c,LDL-c).

SECONDARY OUTCOMES:
Quality of life of diabetic patients and this will be evaluated by using Quality of Life Questionnaire (Short Form 36 questions (SF-36)) . | Two months
  The effect of Rutin and vitamin C combination on quality of life of diabetic patients before and after treatment for 8 weeks and this will be evaluated by using Quality of Life Questionnaire (Short Form 36 questions (SF-36)) .

CONTACTS AND LOCATIONS:
Overall Officials: sara R Ragheb, master, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Ragheb SR, El Wakeel LM, Nasr MS, Sabri NA. Impact of Rutin and Vitamin C combination on oxidative stress and glycemic control in patients with type 2 diabetes. Clin Nutr ESPEN. 2020 Feb;35:128-135. doi: 10.1016/j.clnesp.2019.10.015. Epub 2019 Nov 14. PMID 31987106